CLINICAL TRIAL: NCT02152540
Title: Repetitive Transcranial Magnetic Stimulation to Improve Cognitive Function in TBI
Brief Title: rTMS to Improve Cognitive Function in TBI
Acronym: rTMSTBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N1416-P; RX13-011 (Other Grant/Funding Number: VA Rehab)
Record Dates: First submitted 2014-05-22; First posted 2014-06-02 (Estimated); Results first posted 2019-05-07 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2020-12

CONDITIONS: Traumatic Brain Injury
Keywords: TBI; Transcranial Magnetic Stimulation, Repetitive; magnetic resonance imaging functional; Quality of life; Executive Function; Veterans
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- ACTIVE rTMS (Experimental): Those receiving experimental treatment will receive 20 sessions of rTMS. The treatment will be delivered by trained medical personnel.
  Interventions: Device: rTMS
- Sham rTMS (Placebo Comparator): Those receiving the sham rTMS will receive 20 sessions of sham rTMS. The treatment will be delivered by trained medical personnel.
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: rTMS — Repetitive Transcranial Magnetic Stimulation
  Arms: ACTIVE rTMS
Device: Sham rTMS — Placebo Device that simulates active rTMS treatment
  Arms: Sham rTMS

SUMMARY:
This project will study 40 Veterans identified with symptoms understood to characterize mild to moderate Traumatic Brain Injury (TBI) including Post Traumatic Stress Disorder (PTSD). Following screening and informed consent, Veterans will be randomly assigned to treatment with repetitive Transcranial Magnetic Stimulation (rTMS) or sham rTMS (placebo). Additional examinations will compare brain imaging (structural and functional MRI scans at rest) across participants at baseline, after acute rTMS treatment, and at 6 month followup. The VA population differs significantly from populations that have been included in prior trials of rTMS for many conditions such as depression, chronic pain, and PTSD. Many returning Operation Enduring Freedom (OEF)/Operation Iraqi Freedom (OIF) personnel and Veterans with concussion histories report cognitive problems, such as impaired attention, verbal fluency, poor planning, reduced working memory, and mental flexibility. The investigators hope to show the efficacy and durability of rTMS in treating these symptoms safely in Veterans with co-morbidities.

DETAILED DESCRIPTION:
The goal of the present study is to evaluate the efficacy and durability of benefits of repetitive Transcranial Magnetic Stimulation (rTMS) as a promising non-invasive therapeutic treatment for executive function deficits reported in Veterans with mild to moderate Traumatic Brain Injury (TBI) patients. Although much progress has been made towards understanding the various deficits following TBI, progress has yet to be made towards identifying and assessing therapeutic treatment options that are responsive to TBI symptoms. Many returning OEF/OIF Veterans with concussion histories report cognitive symptoms that may last for months or years, and affect every day function. Symptoms faced by Veterans with mild to moderate TBI include executive function deficits such as impaired attention (including shifting sets), verbal fluency, poor planning, reduced working memory, and mental flexibility. The primary objective is to assess the efficacy of rTMS in Veterans with mild to moderate TBI in improving executive functioning.

A recent VA study reported improvements in PTSD and related symptoms in Veterans with PTSD who received rTMS (Watts et al., 2012). Repetitive TMS is a method of delivering therapeutic, non-invasive brain stimulation that is currently being used at the VA Palo Alto and Stanford University in a number of clinical trials.

For this pilot study the investigators propose to enroll 40 Veterans diagnosed with mild to moderate TBI (age range 20-65). Inclusion Criteria: mild and moderate TBI will be defined as: post-traumatic amnesia (PTA < 1 day for mild; 1 day> x < 7days for moderate). Because of the extensively documented co-occurrence of TBI with PTSD, (Veterans with TBI with and without PTSD will be enrolled). PTSD will be assessed using standard clinical measures. Exclusionary criteria: patients will be screened for TMS and MRI safety. The duration of the study will be two years, with a 1.5 year enrollment period, and a final half-year of follow-up completion. Following a preliminary telephone screen, Veterans will be scheduled for onsite informed consent, screening, and baseline assessments. Using an electronic randomization form, participants will be enrolled into two groups: active rTMS or sham rTMS. As this is a double blind placebo controlled study, only the subject ID number is provided to the nurse administrating the rTMS treatment. After randomization, the rTMS nurse will test the motor threshold (MT) for rTMS. Each participant will be in the trial for a total of approximately (28) weeks: 1-2 weeks screening, (2) weeks acute treatment phase (including MRI pre and post rTMS) and 24 weeks (6 month) follow-up phase (with MRI, neuropsychological testing and self-report measures). Left Dorsolateral Prefrontal Cortex (DLPFC) will be the stimulation site as it is shown to be affective in treatment of depression and approved by FDA. All participants will receive a minimum of 20 treatments before being evaluated for change in executive function (primary outcome measure).

The primary hypothesis is that Veterans receiving active rTMS will show improvement more than sham treated Veterans in (performance between baseline and last assessment of >1 SD on either the Trail Making Test part B, Delis-Kaplan Executive Function System [D-KEFS] Verbal Fluency and/or D-KEFS Color-Word Interference Test). Additional analysis will include: Sustained Improvement on executive function composite score; secondary consequences of TBI scores on Quality of Life (QOL) scale, moderators of response such as age, severity of symptoms at baseline, type of comorbidity (e.g., PTSD); and, functional brain activity changes with rTMS treatment. This pilot study will be one of the first to demonstrate rTMS as a treatment for executive function deficit in Veterans with mild to moderate TBI. Additionally, it would also report on the efficacy of using functional MRI (fMRI) as a biomarker to capture this improvement in executive function.

ELIGIBILITY:
Inclusion Criteria:

* Veteran of any combat era
* Both Genders
* 20-65years
* (History of (Post Traumatic Amnesia < 1 day for mild TBI; 1 day> x < 7days for moderate TBI))
* Ability to obtain a Motor Threshold (MT) will be determined during the screening process.
* If on a psychotropic medication regimen, that regimen will be stable for at least 4 weeks prior to entry to the study and patient will be willing to remain on a stable regimen during the acute treatment phase.
* Has an adequately stable condition and environment to enable attendance at scheduled clinic visits.
* For female participants, agrees to use one of the following acceptable methods of birth control: abstinence, oral contraceptive; Norplant
* Able to read, verbalize understanding, and voluntarily sign the Informed Consent Form prior to participating in any study-specific procedures or assessments.

Exclusion Criteria:

* Pregnant or lactating female.
* Unable to be safely withdraw, at least two-weeks prior to treatment commencement, from medications that substantially increase the risk of having seizures
* Have a cardiac pacemaker or a cochlear implant
* Have an implanted device (deep brain stimulation) or metal in the brain (see standard MRI exclusion criteria including metal screening section in telephone screen, Appendix A).
* Have a mass lesion, cerebral infarct or other active central nervous system (CNS) disease, including a seizure disorder.
* Known current psychosis as determined by DSM-IV coding in chart (Axis I, psychotic disorder, schizophrenia) or a history of a non-mood psychotic disorder.
* Diagnosis of Bipolar Affective Disorder (as determined by chart review and intake interview)
* Current amnesic disorders, dementia, mini mental state examination (MMSE) 24 or delirium.
* Current substance abuse (not including caffeine or nicotine) as determined by positive toxicology screen, or by history via AUDIT, within 3 months prior to screening
* Prior history of seizures
* Severe TBI or open head injury
* TBI within last two months or in acute stage
* Participation in another concurrent clinical trial
* Patients with prior exposure to rTMS/ECT
* Active current suicidal intent or plan. Patient at risk for suicide will be required to establish a written safety plan involving their primary psychiatrist and the treatment team before entering the clinical trial

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maheen M Adamson, PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Click here for more information about this study: Repetitive Transcranial Magnetic Stimulation to Improve Cognitive Function in TBI — http://www.warrelatedillness.va.gov/

RESULTS

PARTICIPANT FLOW:
Groups:
- rTMS: Those receiving experimental treatment will receive 20 sessions of rTMS. The treatment will be delivered by trained medical personnel.
  rTMS: Repetitive Transcranial Magnetic Stimulation
Period: Overall Study
Arm/Group | rTMS | Sham rTMS
Started | 17 | 16
Completed | 17 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rTMS | Sham rTMS | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 16 | 33
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (13.3) | 39.4 (11.9) | 44.4 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 0 | 5
  Male | 12 | 16 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 2 | 3
  White | 11 | 8 | 19
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 16 | 33
Trails B T-score [Mean (Standard Deviation); unit: T-score] — T-score for Trails B task measuring Executive Function: minimum of 0 and a maximum of 100
  T-score | 52.1 (8.2) | 45.3 (14.9) | 48.7 (11.6)

OUTCOME MEASURES:

1. Primary Outcome: Trail Making Test Part B
Description: The primary hypothesis is that Veterans receiving active rTMS will show improvement more than sham treated Veterans in performance between baseline and last assessment of >1 SD on the Trail Making Test part B. This test is known for its accurate assessment of executive function in mild and moderate TBI.
  The TMT is a timed test and the goal is to complete the test as accurately and as quickly as possible. Raw scores are reported in seconds to complete the test. For Part B, an average score is 75 seconds and a deficient score is greater than 273 seconds.
  The present study reports T-scores, which can range from a minimum of 0 and a maximum of 100. The higher the T- score achieved by a participant, the better the performance, indicating a higher level of functioning.
Time Frame: Baseline (up to two weeks after screening visit); Post-Treatment (2 weeks from end of Baseline up to one month from entering the study but always the day of last treatment)
Measure: Mean (Standard Error); unit: T-score
Arm/Group | rTMS | Sham rTMS
Number analyzed (Participants) | 17 | 16
T-score
  Baseline | 52.1 (14.9) | 45.3 (13.7)
  post-treatment | 52.9 (8.2) | 50.8 (10.3)

2. Secondary Outcome: Sustained Improvement on Executive Function
Description: Hypothesis: At the end of the 6 month post treatment followup TBI patients who received rTMS would be more likely to continue to have greater "executive function improvement" on Trail making test part B than patients who received Sham rTMS.
  Outcome measures Description: Trials B T-score range 0-75; higher scores indicate better performance on T-score
Time Frame: 6-month post treatment follow up
Population: All 25 Veterans met criteria for mild and moderate TBI based on the VA/DOD definition and a neurologist's physical exam.
Measure: Mean (Standard Deviation); unit: T-score
Groups:
- ACTIVE rTMS: Those receiving experimental treatment will receive 20 sessions of rTMS. The treatment will be delivered by trained medical personnel.
  rTMS: Repetitive Transcranial Magnetic Stimulation
  n = 12
- Sham rTMS: Those receiving the sham rTMS will receive 20 sessions of sham rTMS. The treatment will be delivered by trained medical personnel.
  Sham rTMS: Placebo Device that simulates active rTMS treatment
  n = 13
Arm/Group | ACTIVE rTMS | Sham rTMS
Number analyzed (Participants) | 12 | 13
T-score | 51.3 (5.4) | 51.2 (12.9)

3. Secondary Outcome: Change in Quality of Life (QOL) Scale
Description: The Veterans RAND 36 Item Health Survey (VR-36©) is a brief, generic, multi-use, self-administered health surveys comprised of 36 items The instruments are primarily used to measure health-related quality of life, to estimate disease burden and to evaluate disease-specific impact on general and selected populations. The items on the questionnaire correspond to eight principal health domains including general health perceptions, physical functioning, role limitations due to physical and emotional problems, bodily pain, energy-fatigue , social functioning and mental health. higher scores mean better health and depicted in percentages. This scale would show significantly greater improvement in patients with mild to moderate TBI who received rTMS treatment.
  Outcome variable description: Scores for each domain are from 0-100 with a higher score defining a more favorable health outcome.
Time Frame: baseline and immediately post treatment (~two weeks)
Population: All 33 Veterans met criteria for mild and moderate TBI based on the VA/DOD definition and a neurologist's physical exam. All patients went through baseline testing that collected demographic (including military history etc.), neuropsychological and self-report questionnaires for health problems.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | rTMS | Sham rTMS
Number analyzed (Participants) | 17 | 16
score on a scale | 59.0 (23.1) | 58.1 (25.7)

4. Secondary Outcome: Moderators of Response: PTSD Score
Description: Moderators of response Post Traumatic Stress Disorder (PTSD) as measured by PTSD Checklist- Military. The Score range is 17-85; higher scores indicate more severe symptoms.
Time Frame: Baseline only
Population: All 33 Veterans met criteria for mild and moderate TBI based on the VA/DOD definition and a neurologist's physical exam. All patients went through baseline testing that collected demographic (including military history etc.), neuropsychological and self-report questionnaires for health problems including PTSD. Mean Scores for PTSD Checklist are reported here between Sham and Active rTMS groups.
Measure: Mean (Standard Deviation); unit: score on the scale
Groups:
- ACTIVE rTMS: Those receiving experimental treatment will receive 20 sessions of rTMS.
  rTMS: Repetitive Transcranial Magnetic Stimulation
  Here we report the results where we adjusted for PTSD to predict Trails B performance
- Sham rTMS: Those receiving the sham rTMS will receive 20 sessions of sham rTMS. The treatment will be delivered by trained medical personnel.
  Sham rTMS: Placebo Device that simulates active rTMS treatment
  Here we report the results where we adjusted for PTSD to predict Trails B performance.
Arm/Group | ACTIVE rTMS | Sham rTMS
Number analyzed (Participants) | 17 | 16
score on the scale | 41.8 (19.4) | 38.7 (11.8)

5. Secondary Outcome: Treatment Induced Change in Functional Connectivity
Description: Each participant went under an MRI scan at post treatment (2 weeks) and 6-months. Functional MRI measures the Blood Oxygen Level Dependent (BOLD) signal in the brain and it can change with this brain stimulation. One common way to address this change or response to treatment is to measure the connectivity between BOLD signal of a network, such as the established default mode network, with the stimulation site. This is provided as a correlation value between the two points- and the strength of correlation is used for each participant at each time point to see if any change has occurred due to stimulation (active vs. placebo). Beta Values are provided below.
Time Frame: post treatment (2 weeks) and 6-months
Population: We only analyzed 12 participants MRI scans in each group (Active and sham) because some data was lost due to MRI server issue. We are providing Beta scores means and stand below that are from the FMRI connectivity analysis from post treatment to 6-months in Sham and Active groups.
Measure: Mean (Standard Error); unit: beta coefficient
Groups:
- Sham rTMS: Those receiving the sham rTMS will receive 20 sessions of sham rTMS. The treatment will be delivered by trained medical personnel.
  Sham rTMS: Placebo Device that simulates active rTMS treatment
  n = 12
Arm/Group | ACTIVE rTMS | Sham rTMS
Number analyzed (Participants) | 12 | 12
beta coefficient | -0.81 (0.12) | 0.34 (0.15)

6. Secondary Outcome: Change in a Mediator of Response: Brain Derived Neurotrophic Factor (BDNF)
Description: Mediator of response to treatment: to establish a preliminary understanding of the underlying mechanisms related to rTMS modulation of synaptic repair in TBI we will also look at the change from baseline and post treatment in brain-derived neurotrophic factor (BDNF) samples in our population.
  Outcome Measure description: mean of BDNF/ProBDNF ratio measured in blood (ng/ml) will be provided
Time Frame: baseline and post treatment (2 weeks)
Population: We present the mean ratio of Brain Derived Neurotrophic Factor (BDNF)/Pro-BDNF in Active vs. Sham groups from baseline to post treatment
Measure: Mean (Standard Deviation); unit: ratio of BDNF/Pro-BDNF
Groups:
- ACTIVE rTMS: Those receiving experimental treatment will receive 20 sessions of rTMS. The treatment will be delivered by trained medical personnel.
  rTMS: Repetitive Transcranial Magnetic Stimulation
  n = 17
- Sham rTMS: Those receiving the sham rTMS will receive 20 sessions of sham rTMS. The treatment will be delivered by trained medical personnel.
  Sham rTMS: Placebo Device that simulates active rTMS treatment
  n = 16
Arm/Group | ACTIVE rTMS | Sham rTMS
Number analyzed (Participants) | 17 | 16
ratio of BDNF/Pro-BDNF | -0.31 (3.02) | 0.25 (3.10)

ADVERSE EVENTS:
Time Frame: 6 months (from first rTMS treatment to 6 month follow up)
Arm/Group | rTMS | Sham rTMS
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 6/17 | 0/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rTMS (N=17) | Sham rTMS (N=16)
Pain behind R eye for 5 minutes (Eye disorders) | 1 (1) | 0 (0)
Sensation of decreased hearing acuity, pt realized was more "aware" of hearing (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Pressure behind eyes and headache starting after baseline MRI, resolved in 3 days during first treat (Eye disorders) | 1 (1) | 0 (0)
Exacerbation of low back pain, resolved in 3 days w medication (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Stimulation-induced eye lid and facial twitching due to improper coil positioning, resolved in secs (Eye disorders) | 1 (1) | 0 (0)
Headache after treatment, resolved same day w/out treatment (Vascular disorders) | 1 (1) | 0 (0)
hematoma at surgery site after parathyroidectomy, unrelated to study participation (Endocrine disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2018-12-11): https://cdn.clinicaltrials.gov/large-docs/40/NCT02152540/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2018-12-11): https://cdn.clinicaltrials.gov/large-docs/40/NCT02152540/SAP_001.pdf